CLINICAL TRIAL: NCT05010252
Title: The Effect of Cycled Light on the Physiological and Visual Development of Premature Infants and the Mother's Sleep and Quality of Life
Brief Title: The Effect of Cycled Light on Premature Infants and Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taiwan Nurses Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202012022RIND
Record Dates: First submitted 2021-07-01; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Preterm Infant Development; Retinopathy of Prematurity; Sleep Quality; Quality of Life
Keywords: Cycled light; retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycled Light (Experimental): It is planned to be in the Neonatal Intermediate Care Nursery, National Taiwan University Children's Hospital, and the subjects are premature babies over 32 weeks old. Divided into two groups of light intervention group and control group, longitudinal tracking intervention effect and six-weeks and three-months delay effect.
  Interventions: Behavioral: Cycled light Experimental
- Dim light (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Cycled light Experimental — The preliminary plan of this study is to carry out empirical evidence and expert advice to confirm precise lighting and develop care intervention strategies for preterm infants based on evidence. It is planned to be in the Neonatal Intermediate Care Nursery, National Taiwan University Children's Hospital, and the subjects are premature babies born 32 weeks old. Divided into two groups of light intervention group and control group, longitudinal tracking intervention effect and six-weeks and three-months delay effect.
  Other Names: Control group
  Arms: Cycled Light

SUMMARY:
Irregular lighting and lack of light in premature infants will affect their health, produce negative effects such as physiological and visual development, and also affect the mother's sleep and quality of life. This study is to verify the effect and delay effect of two-week premature infants' light intervention on their physiological indicators and visual development, mother's sleep quality and quality of life.

It is planned to be in the Neonatal Moderate to Severe Ward of National Taiwan University Children's Hospital, and the subjects are premature babies born 32 weeks old. Divided into two groups of light intervention group and control group, longitudinal tracking intervention effect and six-week and three-month delay effect.

DETAILED DESCRIPTION:
Background Dim, irregular lighting and lack of periodic light in the care environment for premature babies in Taiwan are currently common conditions. Irregular lighting and lack of light in premature infants will affect their health, produce negative effects such as physiological and visual development, and also affect the mother's sleep and quality of life.

Purpose To verify the effect and delay effect of two-week premature infants' light intervention on their physiological indicators and visual development, mother's sleep quality and quality of life.

Methods The preliminary plan of this study is to carry out empirical evidence and expert advice to confirm precise lighting and develop care intervention strategies for preterm infants based on evidence. It is planned to be in the Neonatal Moderate to Severe Ward of National Taiwan University Children's Hospital, and the subjects are premature babies born 32 weeks old. Divided into two groups of light intervention group and control group, longitudinal tracking intervention effect and six-week and three-month delay effect.

ELIGIBILITY:
Inclusion criteria: (1) Premature infants over 32 weeks old, (2) Stable physiological conditions.

Exclusion criteria: (1) taking drugs that may interfere with sleep, (2) suffering from retinopathy (ROP) stage 3 or higher, (3) suffering from intracranial hemorrhage, grade 3 or higher, (4) suffering from upper limb injury or movement disorders, (5) The family has alcohol and drug abuse problems, (6) currently using respirators.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Changes in mean daily Heart Rate during the intervention | up to 42 days
  This is to evaluate the effect of cycled light intervention on Heart Rate (beats/min) in preterm infants. Heart Rate is recorded every 5 minutes. Take the daily average of the Heart Rate, and then analyze its daily change before discharge. The intervention time is after the parents of premature infants agree to participate and before premature infants are discharged from the hospital.
Changes in mean Respiratory Rate during the intervention | up to 42 days
  This is to evaluate the effect of cycled light intervention on Respiratory Rate (breaths/min) in preterm infants. Respiratory Rate is recorded every 5 minutes. Take the daily average of the Respiratory Rate, and then analyze its daily change before discharge. The intervention time is after the parents of premature infants agree to participate and before premature infants are discharged from the hospital.
Changes in mean daily oxygen saturation during the intervention | up to 42 days
  This is to evaluate the effect of cycled light intervention on oxygen saturation SpO2 (%) in preterm infants. Oxygen saturation SpO2 is recorded every 5 minutes. Take the daily average of the oxygen saturation SpO2, and then analyze its daily change before discharge. The intervention time is after the parents of premature infants agree to participate and before premature infants are discharged from the hospital.
Changes in daily body weight during the intervention | up to 42 days
  This is to evaluate the effect of cycled light intervention on body weight (kilograms) in preterm infants. Body weight is recorded every day during hospital stay after intervention, and then we analyze its daily change before discharge. The intervention time is after the parents of premature infants agree to participate and before premature infants are discharged from the hospital.
Mother's sleep quality assessed by the CPSQI [followed by its scale information in the Description] | O1 (before intervention); O2 (at the sixth week after birth); O3 (at the third month after birth)
  Measured by Pittsburgh Sleep Quality Index (CPSQI). Effect of light intervention in premature infants on mother's sleep quality. Data will be collected for the first time (O1) before the experiment, post-test (O2) will be performed six weeks after the intervention, and post-test (O3) will be performed three months after the intervention.
Mother's quality of life assessed by the WHOQoL-BREF [followed by its scale information in the Description] | O1 (before intervention); O2 (at the sixth week after birth); O3 (at the third month after birth)
  The measurement was conducted by the World Health Organization Quality of Life Brief (WHOQoL-BREF) questionnaire. Effect of light intervention in premature infants on mother's quality of life. Data will be collected for the first time (O1) before the experiment, post-test (O2) will be performed six weeks after the intervention, and post-test (O3) will be performed three months after the intervention.

SECONDARY OUTCOMES:
Length of stay in days | at hospital discharge from 0 to 42 days
  Effect of light intervention in premature infants on length of stay.
Weight change | O1 (before intervention); O2 (at the sixth week after birth); O3 (at the third month after birth)
  Effect of light intervention in premature infants on weight (kilograms).
Severity of retinopathy of prematurity (ROP) | O1 (before intervention); O2 (at the sixth week after birth); O3 (at the third month after birth)
  ROP is described by its location in the eye (the zone), by the severity of the disease (the stage) and by the appearance of the retinal vessels (plus disease). The first stage of ROP is a demarcation line that separates normal from premature retina. Stage 2 is a ridge which has height and width. Stage 3 is the growth of fragile new abnormal blood vessels. The severity of ROP is judged by the doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Shin Fen Lee, Head Nurse, Principal Investigator — National Taiwan University Children Hospital; Ciao-Lin Ho, PhD, Principal Investigator — Second Degree Bachelor of Science in Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174